CLINICAL TRIAL: NCT02676817
Title: Probe-based Confocal Laser Endomicroscopy for Assessment of Mucosal Healing in Ulcerative Colitis: Development and Validation of the ENHANCE Score
Brief Title: Confocal Laser Endomicroscopy for Assessment of Mucosal Healing in Ulcerative Colitis
Acronym: ENHANCE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, RAHMI Gabriel, Medical Doctor, European Georges Pompidou Hospital
Other Study IDs: 2014-A00990-47
Record Dates: First submitted 2015-08-14; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Colitis, Ulcerative
Keywords: colitis; endoscopy
MeSH Terms: conditions — Colitis, Ulcerative; Colitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colonic biopsies wre taken during colonoscopy in order to assess the histological inflammation and to correlate the result with pCLE description.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Group 1 (n=70) = UC in remission regardless of the medication that allowed remission nor taken by the patient (Mayo' sub-score 0 or 1) and who require colonoscopy regardless of the study according to current guidelines (screening for dysplasia, monitoring during treatment etc).
- Group 2: Group 2 (n=30) = Active UC (Mayo' sub-score 2 or 3) requiring adalimumab and for whom a rectosigmoidoscopy will be performed 8 to 12 weeks after starting therapy, according to current French guidelines and routine practice. Eight weeks after the treatment is the minimum time necessary to evaluate the effects of this treatment according the current practice in France. Then, investigators chose in our study to assess the effects in the group 2 at 8 weeks. All the 30 patients in group 2 will receive adalimumab and they will be anti-TNF naïve patients.

SUMMARY:
The aim of the study is to construct and validate an endomicroscopic score correlated with microscopic inflammation activity in patients with UC.

Probe-based confocal laser endomicroscopy (pCLE) is a new endoscopic imaging modality, which offers the possibility to perform in vivo mucosal microscopic analysis in real time during endoscopy.

Primary Objectives : Development and validation of a UC endomicroscopic score, after correlation between pCLE data and histological data using the Geboes' score as a gold standard during ulcerative colitis.

Secondary Objectives:

* Identify predictive factors for the response to adalimumab.
* Identify predictive factors for recurrence in patients with UC in remission (Mayo score 0 or 1).
* Safety of the pCLE procedure

DETAILED DESCRIPTION:
Informed consent will be obtained before colonoscopy that includes the known risks and benefits related to the procedure according to the standard protocol of the physician and institution.

A separate informed consent document to participate in the study specific to the approach, technology will be executed.

1. Operator's training before the beginning of the study

   Thirty short pCLE video sequences will be sent to each investigator. Video sequence contains pCLE images of mucosal inflammation in a patient with UC. For each video the correlation with histology is known. The investigator will have to recognize the different pCLE inflammation criteria (Annex 2) and a 90% correct response rate will be required.
2. Endoscopic procedures

MACROSCOPIC examination: colonoscopy

Bowel preparation according to standard protocol was used for colonoscopy. During the colonoscopy, the rectal and colonic mucosal will be analysed with high resolution white light (with or without virtual chromoendoscopy). Before pCLE examination and according to current guidelines, targeted biopsies will be taken in every suspected area of dysplasia for specific histological examination.

MICROSCOPIC examination: pCLE (Cellvizio)

pCLE examination will be done after intravenous injection of fluoresceine (2.5 ml), with the monitoring of cardiovascular and respiratory functions. Three defined area will be analysed: right colon, left colon (40cm from the anus) and the rectum (10cm). Real time analysis and re-reading after the colonoscopy will be done for the video sequences recording during the procedure. A double-blind analysis for each video sequence will be done by two experienced endoscopists.

Rectal and colonic biopsies

For each location (right colon, left colon and rectum), 4 macroscopic area will be indentified (anterior, posterior, left and right), recorded (endoscopic images) and the mucosal inflammation will be scored according to the Mayo's and UCEIS classifications. Then, the probe using for the pCLE procedure will be applied on these 4 different areas and video sequences will be recorded ("optical biopsies"). At the end of the procedure, biopsies will be taken from each area. Each biopsy will have a registration number and the corresponding pCLE video sequence will be specified.

For each location (right colon, left colon, rectum), the final score of inflammation (macroscopic or microscopic) will be define by the higher score recorded in the 4 areas (anterior, posterior, left and righ).

Sensibility to change

For the patients with active UC in group 2 (Mayo' sub-score 2 or 3), a rectosigmoidoscopy should be performed 8 weeks after starting therapy, according to current french guidelines. In order to compare the pCLE examination before and after adalimumab therapy in the group 2, each area will be identified with a submucosal injection of Indian ink.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of UC established at least for three months, according to the Lennard-Jones' criteria. Two sub-groups will be studied as follows;

  * Group 1 (n=70) = UC in remission regardless of the medication that allowed remission nor taken by the patient (Mayo' sub-score 0 or 1) and who require colonoscopy regardless of the study according to current guidelines (screening for dysplasia, monitoring during treatment etc).
  * Group 2 (n=30) = Active UC (Mayo' sub-score 2 or 3) requiring adalimumab and for whom a rectosigmoidoscopy should be performed 8 weeks after starting therapy, according to current french guidelines. Eight weeks after the treatment is the minimum time necessary to evaluate the effects of this treatment according the current practice in France. Then, investigators chose in our study to assess the effects in the group 2 at 8 weeks. All the 30 patients in group 2 will receive adalimumab and they will be treatment-naïve patients.
* Informed consent obtained from the patient

Exclusion Criteria:

* Allergy to fluorescein
* Pregnancy
* Refusal to participate to the study or inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with UC who need control coloscopy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Inflammation assessment by pCLE videos and standard histology | 6 months
  Inflammation will be present if ONE or MORE of the following criteria will be showed by the pCLE examination (the number of criteria will be defined "a posteriori" after comparison with the histological results):
  * crypt: : number (0-10), size (10 to 200 micrometers), distance between 2 crypts (increase or normal)
  * cells : number (0 to 50), color (white or black)
  * vessels : number, diamter (> or < 20 micrometers)
  * fluoresceine leakage (yes or no)

SECONDARY OUTCOMES:
Changes in pCLE criteria after adalimumab and safety of pCLE | 6 or 8 weeks
  Inflammation will be present if ONE or MORE of the following criteria will be showed by the pCLE examination (the number of criteria will be defined "a posteriori" after comparison with the histological results):
  * crypt: : number (0-10), size (10 to 200 micrometers), distance between 2 crypts (increase or normal)
  * cells : number (0 to 50), color (white or black)
  * vessels : number, diamter (> or < 20 micrometers)
  * fluoresceine leakage (yes or no) pCLE safety (intravenous fluoresceine): cardiological trouble: yes or no allergy (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: gabriel rahmi, MD, Principal Investigator — European Georges Pompidou Hospital
Locations (1):
- Hôpital Europeén Georges Pompidou, Paris, France